CLINICAL TRIAL: NCT05855772
Title: Effect of Extracorporeal Shockwave Therapy Before Postural Correction Exercise on EMG Ratio, CVA, PPT, and NDI in Adults With Forward Head Posture
Brief Title: Effect of Extracorporeal Shockwave Therapy Before Postural Correction Exercise in Adults With Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Soyeon Kim, Physical Therapist, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYU 2023-02-007-001
Record Dates: First submitted 2023-04-26; First posted 2023-05-11 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain; Extracorporeal Shock Waves Therapy; Exercise Program
Keywords: Forward head posture; Extracorporeal shock waves; Posture Corrective Exercise Program; Trigger point; Upper trapezius; Serratus anterior; Middle trapezius; lower trapezius; Musculoskeletal Pain
MeSH Terms: conditions — Neck Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock waves therapy[ESWT] + posture corrective exercise programs[PCEP] (Experimental): Before proceeding with the exercise, apply a radial-type Extracorporeal shock waves. This applies to the main muscles with TrP, the upper trapezius and Leavator scapulae muscle. It is conducted twice a week at 1000 impulse, 60 mJ/m (2), and 5 Hz frequencies. In addition, a posture correction exercise program will be conducted along with ESWT. Muscles such as weakened deep neck flexors, middle trapezius muscles, lower trapezius muscles, and serratus anterior muscles will undergo strengthening exercises, while muscles such as shortened and overactive upper trapezius muscle, Leavator scapulae muscle, and sternocleidomastoid muscle will apply relaxation stretching. This will be conducted privately at home by providing exercise leaflets, and will be conducted for a total of four weeks with a 30-minute program three times a week.
  Interventions: Device: Extracorporeal shock waves; Behavioral: Posture Correction Exercise Program
- posture corrective exercise programs[PCEP] (Active Comparator): Only posture correction exercise programs are conducted. Muscles such as weakened deep neck flexors, middle trapezius muscles, lower trapezius muscles, and serratus anterior muscles will undergo strengthening exercises, while muscles such as shortened and overactive upper trapezius muscle, Leavator scapulae muscle, and sternocleidomastoid muscle will apply relaxation stretching. This will be conducted privately at home by providing exercise leaflets, and will be conducted for a total of four weeks with a 30-minute program three times a week.
  Interventions: Behavioral: Posture Correction Exercise Program

INTERVENTIONS:
Device: Extracorporeal shock waves — Extracorporeal shock waves are non-invasive and simple treatments that are easy to apply to a wide surface and have fewer side effects with low intensity. In addition, there is an advantage of improving blood circulation through an increase in reactive blood flow and creation of new blood vessels.
  Other Names: ESWT
  Arms: Extracorporeal shock waves therapy[ESWT] + posture corrective exercise programs[PCEP]
Behavioral: Posture Correction Exercise Program — The exercise program mainly consists of stretching and muscle strengthening exercises, which have shown improvement effects in terms of head vertebrae and pain. In order to optimize the muscle activity between pairs due to FHP, the selected exercise should focus on providing an appropriate proportion of muscle activity for each other as well as muscle strength.
  Other Names: PCEP

SUMMARY:
Currently, as digital leisure activities increase, more time is spent at home. According to these social trends, it is necessary to establish a program that can safely and effectively perform exercise at home.Therefore, this study assumed that if the trigger point and tension of the upper trapezius are resolved by applying ESWT before implementing the exercise program, it will have a significant effect on pain, functional aspects, and posture improvement. On this account, investigator would like to study the effect of applying ESWT before conducting the exercise program on the muscle activity ratio, craniovertebral angle, pressure pain threshold, and Neck disability index in adults with FHP.

DETAILED DESCRIPTION:
Experimental participants who meet the criteria of the study subjects will be selected, and the experiment will be conducted by coordinating the schedules of the subjects. The experiment will be conducted in an independent space, and the general characteristics of the subjects will be investigated collectively before the experiment. Subjects will take a side photograph from a distance of 265 cm to check the CVA. In addition, the basic value will be obtained by measuring the activity of the UT, MT, LT and SA when the arm is lifted in the direction of the scapula plane, and the pressure pain threshold of the UT Trigger point will be measured using a pain threshold will be measured. In addition, NDI will be self-measured to evaluate neck pain and function. The experiment will be divided into groups that conduct in ESWT and posture correction exercise programs together and groups that conduct only posture correction exercise programs, and the subjects will be randomly assigned to the two groups. After the experiment is completed, the muscle activity, head spine angle, pressure pain threshold, and ranch index measured in advance will be measured again.

ESWT: Radial shock waves will be applied to the main muscles with Trigger points, the Upper trapezius and Levator scapulae muscles. This is conducted twice a week, with 1000impulses, 60mJ/m (2), and 5Hz frequency for a total of four weeks.

Posture Correction Exercise Program: Muscles such as weakened deep neck flexors, middle trapezius, lower trapezius, and serratus anterior muscles will undergo strengthening exercises, while muscles such as shortened and overactive upper trapezius, Levator scapulae, and sternocleidomastoid muscle will apply relaxation stretching. This will be conducted privately at home by providing exercise leaflets, and will be conducted for a total of four weeks with a 30-minute program three times a week.

ELIGIBILITY:
Inclusion Criteria:

* Those with CVA≤53 or less when measuring the Craniovertbral angle through photometric method
* A person who uses a smartphone or computer for an average of 4 hours or more per day
* A person who has not exercised regularly in the past six months

Exclusion Criteria:

* A person who is subject to extracorporeal shock wave contraindication
* A person with a history of fractures or surgery
* A person who is unable to exercise due to medical conditions

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Electromyography | 6weeks
  It will measure muscle activity when the arm is raised in the direction of the scapula plane. Each muscle measured is an upper trapezius, middle trapezius, lower trapezius, and serratus anterior, and the values obtained are to obtain the muscle activity ratio of each of the upper trapezius/lower trapezius, upper trapezius/middle trapezius, upper trapezius/serratus anterior.

SECONDARY OUTCOMES:
Photogrammetry(CVA) | 6weeks
  To check the angle of the head spine, the subjects' profile will be photographed at a distance of 265 centimeters. We would like to measure the angle of the line connecting the migration and cervical spine 7 spinous process in a vertical line to check the change in the angle of the head that comes out forward.
Pressure pain threshold | 6weeks
  It is intended to obtain a quantitative value related to mechanical sensitivity to deep structural pain by applying the metal rod of the pain system vertically to the trigger point area of the upper trapezius.
Neck Disability Index | 6weeks
  We would like to check the difference in the degree of pain and the degree of limitation in daily life due to neck pain by evaluating the items of self-management, lifting objects, reading, headache, concentration, work, driving, sleep and leisure activities as scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Soyeon, Principal Investigator — Sahmyook University
Locations (1):
- Sahmyook university, Seoul, Nowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No